CLINICAL TRIAL: NCT01253135
Title: An Open-label, Randomized, Evaluator-Blinded Study of the Effect of Polymerized Fibrin Applied Topically Once Per Week, on Healing of Induced Thermal Wounds, Versus Weekly Application of White Petrolatum
Brief Title: Study to Determine if Fibrin Affects the Ability of a Wound to Heal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 802-247-09-017
Record Dates: First submitted 2010-11-30; First posted 2010-12-03 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Effect of Test Articles on the Healing of a Wound Artificially Induced by Liquid Nitrogen Spray
Keywords: Fibrin, white petrolatum, wound healing
MeSH Terms: interventions — Fibrin; Petrolatum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): White Petrolatum
  Interventions: Other: White Petrolatum
- Test article (Other): Vehicle (fibrinogen)
  Interventions: Biological: Fibrin

INTERVENTIONS:
Biological: Fibrin — Topical application of fibrinogen spray, followed by thrombin spray
  Arms: Test article
Other: White Petrolatum — Topical application
  Arms: Control

SUMMARY:
The objective of this study is to evaluate the potential inhibitory effects of HP802-247 Vehicle on wound closure (healing), by comparing mean days to closure of superficial (partial-thickness) thermal wounds against similar wounds treated with white petrolatum.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information.
* Are male or female, ≥ 18 years of age, of any race.
* Are willing to attend all required study visits, and to comply with study procedures.
* Meet none of the exclusion criteria (any single exclusion criterion which is met by a potential subject will disqualify that subject from participation in this study.

Exclusion Criteria:

* Have a history of dermatomyositis, systemic sclerosis, scleroderma, Sjögren's syndrome, systemic lupus erythematosus, discoid lupus, Ehler Danlos disease, icthyosis vulgaris, vasculitis, or bleeding disorders (coagulopathies).
* Have any dermatologic disease which may be aggravated or provoked by the wounding procedure, such as Lichen Planus, Psoriasis, or Vitiligo.
* Have Fitzpatrick scale skin type 6 (never sunburns, deeply pigmented).
* Are at risk of keloid or hypertrophic scar formation, based on personal history, family history, or brief skin exam (conducted at the screening visit to look for keloids or hypertrophic scars).
* Have been treated within the last three months for uncontrolled diabetes mellitus, peripheral vascular disease, vitamin C deficiency, connective tissue disorders, or any other disease process that impedes wound healing.
* Are taking concomitant medications at doses which are known to interfere with healing, such as non-steroidal anti-inflammatory drugs, anti-neoplastic drugs, or immunosuppressive drugs.
* Are using topical glycolic acid products, alpha-hydroxy acid products, retinoids, or chemical peel agents in the treatment areas.
* Are using systemic steroids or immunosuppressant agents, or have used these drugs within the past three months.
* The Principal Investigator may declare any subject ineligible for a valid medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Dermatology, University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Vivas A, Fox JD, Baquerizo Nole KL, Maderal AD, Badiavas E, Cargill DI, Slade HB, Feldman SR, Kirsner RS. Cryo-Induced Thermal Wounds: A Human Acute Wound Model. J Drugs Dermatol. 2015 Jul;14(7):734-8. PMID 26151791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a single US investigation site, between February 2, 2011 and July 5, 2011.
Pre-assignment Details: Subjects who met all inclusion/exclusion criteria received paired superficial thermal injuries, one on the ventral aspect of each forearm, using liquid nitrogen. The test article applied to each arm was determined by randomization code. Wound status (closed/open) was assessed by a blinded assessor.
Groups:
- All Participants: The original protocol (Version 1) called for weekly application of HP802-247 Vehicle alone to the appropriate wound and application of White Petrolatum once weekly to the other wound. After enrollment of the first 15 subjects, scabbing was noted over both wounds, making it impossible to determine the day of wound closure. It was conjectured that the wound environment was becoming too dry. Version 1 of the protocol was stopped and it was amended to Version 2, in which White Petrolatum as applied daily to both wounds. On the days that HP802-247 Vehicle was applied, the White Petrolatum was applied 5 min later to allow the fibrin matrix to mature. 25 subjects were enrolled under Version 2. All 40 subjects enrolled in the study were assessed for safety and the 25 subjects enrolled under Version 2 were assessed for wound closure.
Period: Original Protocol
Arm/Group | All Participants
Started | 15
Completed | 0
Not Completed | 15
Not completed — Protocol Amendment | 15
Period: Amended Protocol
Arm/Group | All Participants
Started | 25
Completed | 24
Not Completed | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Population: There were 40 participants in the entire study. Only 25 participants in the amended protocol
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Customized [Mean (Standard Deviation); unit: years]
  Age for all 40 participants | 30.7 (10.2)
  Age for only amended protocol participants | 32.8 (11.3)
Sex/Gender, Customized [Number; unit: participants]
  Male entire study population | 20
  Female entire study population | 20
  Male amended protocol | 13
  Female amended protocol | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 32
  More than one race | 3
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants] — For amended protocol participants
  participants
    Hispanic/Latino | 15
    Non Hispanic/Latino | 10
    Asian | 1
    Black/African American | 3
    White/Caucasian | 18
    Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Time (in Days) to Wound Closure (Healing) Defined as Skin Re-epithelialization, Without Drainage or Dressing Requirements.
Description: The target wounds were evaluated wound status (open/closed).
Time Frame: All thermal wound injury was done on Day 1. Application of test articles started on Day 2. Target wound assessment was performed on Day 3 and Day 5; subsequent assessments were done Monday through Friday for 2 weeks and subjects exited study on Day 22
Population: ITT Populations: Subjects who participated in version 2 of the protocol. Inter-group comparison was done using a paired Prentice-Wilcoxon method, which is applicable to censored data.
Measure: Mean (Standard Deviation); unit: days to wound closure
Groups:
- Control: White Petrolatum
  White Petrolatum: Topical application
  White petrolatum was applied daily to the appropriate wound.
- Test Article: 802-247 Vehicle (fibrinogen)
  Fibrin: Topical application of fibrinogen spray, followed by thrombin spray
  HP802-247 Vehicle (260 µL) was applied to the appropriate wound on days 1, 8, and 15. White petrolatum was applied daily. On days 1, 8,and 15 it was applied 5 min after application of HP802-247 Vehicle, to allow the fibrin matrix to mature.
Arm/Group | Control | Test Article
Number analyzed (Participants) | 25 | 25
days to wound closure | 14.4 (5.5) | 13.3 (3.3)
Statistical Analysis 1: Comparison: Control vs Test Article; Test type: Superiority or Other; p = .3393, Prentice-Wilcoxon test; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.08 to 0.84], Standard Deviation 4.7 — The Confidence Interval was based on a t-distribution

2. Primary Outcome: Median Time (in Days) to Wound Closure (Healing) Defined as Skin Re-epithelialization, Without Drainage or Dressing Requirements.
Description: The target wounds were evaluated wound status (open/closed)
Time Frame: as for outcome 1
Population: ITT Populations: Subjects who participated in version 2 of the protocol. The primary efficacy endpoint was analyzed, using Kaplan-Meier survival analysis, to estimate the median time to wound closure over the 21-day treatment period. Any wound which did not heal by Day 21 was censored in the analysis.
Measure: Median (95% Confidence Interval); unit: days to closure
Arm/Group | Test Article | Control
Number analyzed (Participants) | 25 | 25
days to closure | 12 [11 to 15] | 12 [11 to 15]
Statistical Analysis 1: Comparison: Test Article vs Control; Test type: Superiority or Other; p = .4771, Log Rank; Testing was by a Log Rank test with significance being at P < 0.05

ADVERSE EVENTS:
Time Frame: Safety reporting occurred over the three weeks of the treatment period.
Description: All subjects randomized to treatment were questioned about adverse events and were included in the number of participants assessed for safety. The first assessments at each visit were about changes in general health and concomitant medications and the occurrence of adverse events.
Arm/Group | Control | Test Article
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 18/40 | 18/40
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=40) | Test Article (N=40)
General disorders & administrative site conditions (General disorders) | 3 (6) | 1 (2)
Pain (General disorders) | 2 (3) | 1 (2)
Infections and Infestations (Infections and infestations) | 2 (2) | 2 (2)
Injury, poisoning & procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Musculoskeletal & connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Skin & subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 17 (29) | 17 (29)
Dermatitis (Skin and subcutaneous tissue disorders) | 10 (10) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (18) | 13 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less